CLINICAL TRIAL: NCT04892108
Title: Surgical Treatment of Internal Rectal Prolapse Associated With Obstructed Defecation: Transanal Prolassectomy Versus Laparoscopic Ventral Rectopexy. Randomized Controlled Trial.
Brief Title: Rectal Prolapse With ODS. STARR vs LVR.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Simona Ascanelli, Principal Investigator, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 129/2021/Sper/AOUFe
Record Dates: First submitted 2021-04-11; First posted 2021-05-19 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Rectal Prolapse; Defecation Disorder; Rectocele; Female; Surgery
Keywords: Obstructed defecation syndrome; Transanal rectal prolassectomy; Laparoscopic ventral mesh rectopexy
MeSH Terms: conditions — Rectal Prolapse; Rectocele

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial is designed to compare the outcome of patients with obstructed defecation syndrome (ODS) and rectal prolapse undergoing transanal prolassectomy surgery with mechanical stapler (STARR: stapled transanal rectal resection) versus laparoscopic ventral rectopexy (LVR) surgery, with the aim of evaluating the most appropriate surgical choice. Patients eligible for the study will be randomized on a 1:1 basis to undergo transanal prolassectomy (Group 1: STARR) or laparoscopic ventral rectopexy with mesh placement (Group 2: LVR).
  Randomization will be performed by a randomized list. The assignment sequence will be generated from a random numerical series generated through a computerized list. Randomization will be in blocks of 4. Group assignments will be unknown to those responsible for data collection and those who will be responsible for statistical analysis and clinical evaluation of patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group STARR (Experimental): Patients undergoing transanal prolassectomy with mechanical stapler (STARR: Stapled Trans Anal Rectal Resection) randomly
  Interventions: Procedure: STARR (Stapled Trans Anal Rectal Resection)
- Group LVR (Experimental): Patients undergoing Laparoscopic suspensory correction of rectal prolapse by ventral rectopexy with biological prosthesis (LVR) randomly
  Interventions: Procedure: LVR (Laparoscopic Ventral Rectopexy)

INTERVENTIONS:
Procedure: STARR (Stapled Trans Anal Rectal Resection) — Patients randomly assigned to surgical intervention of STARR (Stapled Trans Anal Rectal Resection)
  Arms: Group STARR
Procedure: LVR (Laparoscopic Ventral Rectopexy) — Patients randomly assigned to surgical intervention of LVR (Laparoscopic Ventral Rectopexy)
  Arms: Group LVR

SUMMARY:
The objective of the study will be to evaluate the clinical and functional outcome of patients with obstructed defecation sndrome (ODS) associated to internal rectal prolapse, treated with transanal prolassectomy (STARR) surgery compared to those treated with laparoscopic ventral rectopexy (LVR).

DETAILED DESCRIPTION:
This randomized controlled trial (single center, prospective, randomized controlled, parallel, and single-blind trial) is designed to compare the outcome of patients with ODS and rectal prolapse undergoing transanal prolapsectomy with mechanical stapler (STARR) versus laparoscopic ventral rectopexy (LVR), with the aim of evaluating the most appropriate surgical choice.

The study will be conducted at the Surgical Unit 2 of the University Hospital of Ferrara, Italy. Patients suffering from rectal prolapse and ODS that will refer to the colorectal and pelvic floor clinic of the University Hospital Ferrara, and eligible for surgery, will be evaluated consecutively after expressing consent to participate in the study by signing an informed consent.

The duration of the study for each patient will be expected to be 48 months with follow-up at 1, 3, 6, 12, 24, 36, and 48 months postoperatively.

Eligible patients will receive information about participating in the trial by their surgeon. Consecutive eligible patients will be randomly assigned to one of two groups with a 1:1 equal allocation ratio.

Patients eligible for the study will be randomized on a 1:1 basis to undergo transanal prolassectomy (Group 1: STARR) or laparoscopic ventral rectopexy with mesh placement (Group 2: LVR).

An independent individual will perform randomization using a software randomization program. Randomization will be performed by a randomized list. The assignment sequence will be generated from a random numerical series generated through a computerized list. Randomization will be in blocks of 4. Group assignments will be unknown to those responsible for data collection and those who will be responsible for statistical analysis and clinical evaluation of patients.

The diagnosis of ODS will be attributed after clinical evaluation at the colorectal clinic and on the basis of the presence of one or more symptoms associated with this disorder, such as to reach a score of 14 and above according to the validated score of ODS of Altomare.

Assessment After recruitment and consent, all patients under study will be asked and collected demographic and clinical information with comorbidities (in particular diabetes, fibromyalgia, depressive disorders, neurological diseases, COPD), parity, previous pelvic surgery, type of surgery, time of hospitalization and any complications (according to Clavien-Dindo classification).

Data concerning the grade of rectoanal prolapse, according with Oxford Classification [20], and rectocele grading will be collected through outpatient proctological evaluation associated with proctoscopy, rectal manometry, and Rx defecography. Colonoscopy will be also performed in every patient to exclude colorectal cancer.

The severity of the ODS will be scored with the Altomare's ODS scoring system. Constipation and fecal incontinence will be measured by obtaining their scores through the administration of validated questionnaires such as the Wexner Constipation score, and the Cleveland Clinic Fecal Incontinence Score (CCFI).

Quality of life will be also evaluated by the patient assessment of constipation quality-of-life (PAC-Qol) questionnaire. The study of eventually associated pelvic distress will be assessed by administering validated questionnaires such as the Pelvic Floor Distress Inventory (PFDI-score, short form) and the Pelvic Floor Impact Questionnaire (PFQI-score, short form).

The scores obtained, as well as the presence of symptoms (fecal incontinence, constipation, or ODS) will be calculated before and after surgery (at 6, 12, 24, 36, and 48 months). All patients will be followed up on an outpatient basis at 7 days, 1 month, 3 months, 6 months, 12 ,24, 36, and 48 months after surgery. Rectal manometry and defecography will be performed after 12 months after surgery.

Surgical intervention All the procedures will be performed by a single surgeon (SA). The LVR technique used for this protocol is as previously described. Subjects randomized to this arm will receive a standard LVR. Briefly, the peritoneum is opened over the right side of the sacral promontory. The mesorectum is dissected and extended in an inverted J-form along the right side. The rectovaginal septum is opened to the pelvic floor. Biologic mesh (Permacol) is sutured to the ventral aspect of the rectum with non-readsorbable stitches. The proximal end of the mesh is fixed on the anterior longitudinal ligament at sacral promontory with nonabsorbable tacks. The incised peritoneum is then closed to over the mesh.

Subjects randomized to STARR arm will undergo a STARR procedure. Briefly, a circular anal dilator is introduced into the rectum. The purse-string anoscope is used to complete the anterior hemi-circumference purse-string suture, about 2-3 cm above the haemorrhoidal apex. A 33-mm circular stapler (Ethicon, ppH01) is opened, inserted until crossing the purse-string which is then tied with a knot. Then the stapler is closed and fired. The same hemi-circumference purse-string suture is performed in the posterior rectal wall. A second application of the stapler on the posterior wall is inserted, closed and fired.

The duration of the study will be 2 years. The study will be conducted in accordance with the principles of Helsinki Declaration, with approval of the medical ethics review board of S. Anna University Hospital. A written informed consent will be obtained from all enrolled patients.

The report will comply with the strengthening the reporting of randomized studies (CONSORT).

ELIGIBILITY:
Inclusion Criteria:

* female gender,
* the presence of rectorectal or rectoanal intussusception as main cause of ODS, confirmed by defecography,
* type of operation performed (STARR or LVR),
* ODS score > 14 [17]
* PACQoL >32 [18]
* ODS symptoms for at least 12 months prior to enrollment
* Failure of at least 6 months of medical therapy

Exclusion Criteria:

* male gender,
* severe fecal incontinence (CCS score>6, Maximum Resting Pressure at rectal manometry < 50 mmHg),
* combined procedures
* previous surgery on rectum or anus for cancer or rectal prolapse, inflammatory bowel disease, other type of surgery to relieve ODS
* pregnancy,
* anismus or dissinergic defecation
* full-thickness prolapse
* stress urinary incontinence associated
* histerocele or cystocele associated (since we usually correct both defects in the same surgical procedure)
* prior pelvic radiotherapy
* slow transit constipation defined as ≤ 2 bowel movements per week,
* any psychiatric diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of different outcomes in relief from ODS after surgery in both groups | 4 years
  In order to evaluate the short- and long-term efficacy of STARR procedure compared to LVR, the percentage of changes in total ODS, PAC-QoL, PFDI, PFQI, Wexner Constipation, the Cleveland Clinic Fecal Incontinence (CCFI) scores between baseline and 6, 12, 24, 36, and 48 months after surgery, were adopted as primary outcome.

SECONDARY OUTCOMES:
short-term postoperative complications (within 30 days after surgery) | 4 years
  short-term postoperative complications (within 30 days after surgery) in the two groups (according to Clavien-Dindo classification)
long-term postoperative complications | 4 years
  Mesh-related complications, rectal stenosis
recurrence or persistence of rectal prolapse | 4 years
  to evaluate recurrence or persistence of rectal prolapse (diagnosed clinically and by postoperative defecography) in both groups, and the need for subsequent corrective surgery
recurrence or persistence of ODS (Obstructed defecation syndrome) | 4 years
  recurrence or persistence of ODS if ODS score > 10
patient satisfaction in terms of pain | 4 years
  patient satisfaction measured by a VAS (Visual Analogue Scale: evaluation of pain in mm: from 0 to 4 mm: no pain; from 5 to 44 mm: little pain; from 45 to 74 mm: moderate pain; from 75 to 100 mm: severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Simona Ascanelli, Principal Investigator — Surgical Department University Hospital Ferrara Italy
Locations (1):
- Surgery 2 Surgical Department, Sant'Anna University Hospital Ferrara, Italy, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hicks CW, Weinstein M, Wakamatsu M, Savitt L, Pulliam S, Bordeianou L. In patients with rectoceles and obstructed defecation syndrome, surgery should be the option of last resort. Surgery. 2014 Apr;155(4):659-67. doi: 10.1016/j.surg.2013.11.013. Epub 2013 Dec 5. PMID 24508117
- [Background] Khaikin M, Wexner SD. Treatment strategies in obstructed defecation and fecal incontinence. World J Gastroenterol. 2006 May 28;12(20):3168-73. doi: 10.3748/wjg.v12.i20.3168. PMID 16718835
- [Background] Rao SS. Dyssynergic defecation. Gastroenterol Clin North Am. 2001 Mar;30(1):97-114. doi: 10.1016/s0889-8553(05)70169-2. PMID 11394039
- [Background] Podzemny V, Pescatori LC, Pescatori M. Management of obstructed defecation. World J Gastroenterol. 2015 Jan 28;21(4):1053-60. doi: 10.3748/wjg.v21.i4.1053. PMID 25632177
- [Background] Gunner CK, Senapati A, Northover JM, Brown SR. Life after PROSPER. What do people do for external rectal prolapse? Colorectal Dis. 2016 Aug;18(8):811-4. doi: 10.1111/codi.13255. PMID 27481719
- [Background] Senapati A, Gray RG, Middleton LJ, Harding J, Hills RK, Armitage NC, Buckley L, Northover JM; PROSPER Collaborative Group. PROSPER: a randomised comparison of surgical treatments for rectal prolapse. Colorectal Dis. 2013 Jul;15(7):858-68. doi: 10.1111/codi.12177. PMID 23461778
- [Background] Emile SH, Elfeki H, Shalaby M, Sakr A, Sileri P, Wexner SD. Perineal resectional procedures for the treatment of complete rectal prolapse: A systematic review of the literature. Int J Surg. 2017 Oct;46:146-154. doi: 10.1016/j.ijsu.2017.09.005. Epub 2017 Sep 7. PMID 28890414
- [Background] van den Esschert JW, van Geloven AA, Vermulst N, Groenedijk AG, de Wit LT, Gerhards MF. Laparoscopic ventral rectopexy for obstructed defecation syndrome. Surg Endosc. 2008 Dec;22(12):2728-32. doi: 10.1007/s00464-008-9771-9. Epub 2008 Mar 5. PMID 18320283
- [Background] Altomare DF, Spazzafumo L, Rinaldi M, Dodi G, Ghiselli R, Piloni V. Set-up and statistical validation of a new scoring system for obstructed defaecation syndrome. Colorectal Dis. 2008 Jan;10(1):84-8. doi: 10.1111/j.1463-1318.2007.01262.x. Epub 2007 Apr 18. PMID 17441968
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Cariou de Vergie L, Venara A, Duchalais E, Frampas E, Lehur PA. Internal rectal prolapse: Definition, assessment and management in 2016. J Visc Surg. 2017 Feb;154(1):21-28. doi: 10.1016/j.jviscsurg.2016.10.004. Epub 2016 Nov 16. PMID 27865742
- [Background] Kluivers KB, Hendriks JC, Shek C, Dietz HP. Pelvic organ prolapse symptoms in relation to POPQ, ordinal stages and ultrasound prolapse assessment. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Sep;19(9):1299-302. doi: 10.1007/s00192-008-0634-7. Epub 2008 May 9. PMID 18465076
- [Background] Agachan F, Chen T, Pfeifer J, Reissman P, Wexner SD. A constipation scoring system to simplify evaluation and management of constipated patients. Dis Colon Rectum. 1996 Jun;39(6):681-5. doi: 10.1007/BF02056950. PMID 8646957
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495
- [Background] Sileri P, Franceschilli L, de Luca E, Lazzaro S, Angelucci GP, Fiaschetti V, Pasecenic C, Gaspari AL. Laparoscopic ventral rectopexy for internal rectal prolapse using biological mesh: postoperative and short-term functional results. J Gastrointest Surg. 2012 Mar;16(3):622-8. doi: 10.1007/s11605-011-1793-2. Epub 2012 Jan 7. PMID 22228202
- [Background] Jayne DG, Schwandner O, Stuto A. Stapled transanal rectal resection for obstructed defecation syndrome: one-year results of the European STARR Registry. Dis Colon Rectum. 2009 Jul;52(7):1205-12; discussion 1212-4. doi: 10.1007/DCR.0b013e3181a9120f. PMID 19571694
- Available data/document: Study Protocol — https://drive.google.com/drive/folders/10w8pl8TztkdTzafLc-M4wRyrHNZI1G-r?usp=sharing
- Available data/document: Statistical Analysis Plan — https://drive.google.com/drive/folders/10w8pl8TztkdTzafLc-M4wRyrHNZI1G-r?usp=sharing
- Available data/document: Informed Consent Form — https://drive.google.com/drive/folders/10w8pl8TztkdTzafLc-M4wRyrHNZI1G-r?usp=sharing